CLINICAL TRIAL: NCT00773344
Title: Phase 1/2 Clinical Trial of the Combination of Trastuzumab (Herceptin) and Tanespimycin
Brief Title: Clinical Trial of the Combination of Trastuzumab (Herceptin) and Tanespimycin in Patients With Solid Tumors and Her2 Positive Metastatic Breast Cancer That Have Previously Failed Herceptin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA200-001; KAG 122
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Solid Tumors; Breast Cancer
Keywords: Solid Tumors (dose escalation/Phase 1); Breast Cancer (recommended dose phase/Phase 2)
MeSH Terms: conditions — Breast Neoplasms | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Tanespimycin

INTERVENTIONS:
Drug: Tanespimycin — Solution, IV, Weekly two hour infusion, 4-cycles until disease progression or DLT
  This is a one-arm study with 4 fixed doses of Tanespimycin (225mg/m2, 300mg/m2, 375mg/m2 and 400mg/m2)
  Other Names: BMS-722782

SUMMARY:
The primary purpose(s) of this study is to determine the highest tolerated dose of tanespimycin and to determine anti-tumor activity (via objective response rate) of tanespimycin in patients with breast cancer who have not previously responded to Herceptin

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* KPS performance status >= 70%
* For the Phase 1 portion of the trial, all patients must have a histologically confirmed solid tumor malignancy. For the Phase 2 portion of the trial, patients must have metastatic breast cancer with HER2 amplification by FISH or 3+ HER2 overexpression by immunohistochemistry ("IHC") Patients may have had either progressive disease within 3 months following last dose of adjuvant treatment with trastuzumab OR progressive disease following initial therapy for metastatic disease with trastuzumab (trastuzumab may have been administered with cytotoxic chemotherapy, hormonal therapy or as single agent.) Patients who have received trastuzumab single agent therapy (without documented progressive disease) followed by trastuzumab combination therapy remain eligible for this study at the time of disease progression. Patients must have measurable disease by RECIST
* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy, must have resolved to NCI CTCAE (v. 3.0) Grade <= 2 (except for alopecia)
* The following laboratory results, within 10 days of KOS-953 administration:
* Hemoglobin >= 8.5 g/dL
* Absolute neutrophils count >= 1.5 x 10*9* /L
* Platelet count >= 75 x 10*9* /L

  * Serum bilirubin <= 2 x ULN
  * AST and ALT <= 2 x ULN
  * Serum creatinine <= 2 x ULN
  * Signed informed consent

Exclusion Criteria:

* Documented hypersensitivity reaction of CTCAE Grade >= 3 to prior therapy containing Cremophor (for those patients who receive the Tanespimycin Injection only) or Herceptin
* Pregnant or breast-feeding women
* Known active CNS metastases
* Except for trastuzumab (Herceptin®) administered between 7-21 days prior to first tanespimycin (KOS-953) administration, administration of any other chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic) within 14 days prior to receipt of study medication. Patients should be 6 weeks from last dose of nitrosourea
* Severe dyspnea at rest caused by complications of advanced malignancy or requiring supplementary oxygen therapy
* Congestive heart failure, or a left ventricular ejection fraction (LVEF) less than 50% assessed by multigated radionuclide angiography scan or echocardiography
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient
* Patients with previous malignancies unless free of recurrence for at least 5 years except cured basal cell carcinoma of the skin, carcinoma-in-situ of either the uterine cervix or urinary bladder, or Stage T1 or T2 prostate cancer whose PSA is < 2 ng/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate (RECIST complete response, or partial response ) confirmed by CT and MRI as the preferred methods for tumor assessments and Chest x-ray is acceptable for pulmonary lesions | Within 28 days prior to the start of treatment with tumor assessments reevaluated every 8 weeks (+/- 4 days)

SECONDARY OUTCOMES:
Kaplan-Meier estimates duration of response and time-to-event variables will be used (time to progression, progression-free survival, time to response, duration of response, time to treatment failure and overall survival) | 3-6 months
Kaplan-Meier estimates duration of response and time-to-event variables will be used (time to progression, progression-free survival, time to response, duration of response, time to treatment failure and overall survival) | 6-12 months
Kaplan-Meier estimates duration of response and time-to-event variables will be used (time to progression, progression-free survival, time to response, duration of response, time to treatment failure and overall survival) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Premiere Oncology Of Arizona, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx